CLINICAL TRIAL: NCT00996086
Title: Risk Stratification and Benefits With Cardiac Resynchronization Therapy
Brief Title: Risk Stratification and Benefits With Cardiac Resynchronization Therapy (CRT)
Acronym: BENEFIT
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Northwestern University (Other); VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CRD 480
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Ventricular Arrhythmias
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — There is a genetic substudy that will evaluate the presence of certain protein markers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CRT device-recipients
  Interventions: Device: CRT device implant

INTERVENTIONS:
Device: CRT device implant — CRT device-recipients

SUMMARY:
This is an observational study to learn which patients benefit from CRT therapy and to track the clinical changes that help identify the risk-level of CRT patients.

DETAILED DESCRIPTION:
The purpose of the study is two-fold. First, to determine if an algorithm can be developed based on pre-implant clinical variables to predict response to CRT-D therapy. Second, the study aims to determine in patients implanted with CRT-D if the combined use of cTnT and BNP can further predict and risk-stratify HF improvement and all-cause mortality. Additionally, novel biochemical markers defining cardiac mortality in high risk patients detected by plasma proteomic analysis in the CRT-D patients will be evaluated.

This study represents a combination of previous CRT studies that evaluated these variables independently. Data from this study will be pooled with data from previous studies to build a more complete picture of CRT therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meets current clinical indications for CRT-D therapy
* Patient is 18 years old or older
* Ability to independently comprehend and complete all QOL questionnaires
* Patient has the ability to perform the 6-minute Hall Walk Test (6-MHW) with the only limiting factor being fatigue or shortness-of-breath
* Ability to provide informed consent for a study and be willing and able to comply with the prescribed follow-up

Exclusion Criteria:

* Inability to successfully implant an intravascular lead and CRT-D device. (i.e. exclude epicardial leads) within 30 days of initial procedure.
* Myocardial infarction in the last 3 weeks
* Unstable angina in the last 3 weeks
* Status 1 classification for cardiac transplantation
* Currently participating in a clinical trial that includes an active treatment arm
* Life expectancy of less than 12 months.
* Recent (within 1 week) administration of Nesiritide™ or inotropes
* Patients in whom revascularization is expected
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo implantation of a market-approved St. Jude Medical CRT defibrillator (CRT-D) and a compatible lead system may be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute hall walk distance between baseline and subsequent follow-up | 12 months
Composite endpoint a. 6-minute hall walk distance b. NYHA Classification c. Quality of Life (Minnesota Living with Heart Failure, DASS, SF-36) | 12 months
The occurrence of either death (all-cause) or first HF hospitalization. | 12 months

SECONDARY OUTCOMES:
Quality of Life | 12 months
Change in echocardiographic variables including: a. Ejection Fraction b. Wall motion score c. Increase in TD velocity d. Yu index | 12 months
Cause-specific mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Kadish, M.D., Principal Investigator — Northwestern University; Alaa Shalaby, M.D., Principal Investigator — VA Pittsburgh Healthcare System
Locations (2):
- United States (2):
  - Touro College, New York, New York
  - Veterans' Adminstration Pittsburgh Healthcare System, Pittsburgh, Pennsylvania